CLINICAL TRIAL: NCT05179174
Title: The Role of Genetic Mutations and of Circulating mRNAs in Uveal Melanoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Antonio Longo, Associate Professor, University of Catania
Other Study IDs: 71/2020/PO
Record Dates: First submitted 2021-09-19; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Uveal Melanoma
Keywords: uveal melanoma; GNA11 mutation; GNAQ mutation; micro RNA
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood from routine sample will be analyzed at the Laboratory of Experimental Oncology of the Department of Biomedical and Biotechnological Sciences, University of Catania, Italy, in order to research the mutations of the GNA11 and GNAQ genes and the following microRNAs: miR - 506-514 cluster, hsamiR - 592 and hsa - miR - 199a - 5p, using the digital PCR droplet system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with uveal melanoma: 51 patients with a diagnosed with uveal melanoma; of both sexes, aging more than 18 years. The exclusion criteria are: a) subjects with autoimmune diseases, tumors, diseases kidney, atherosclerosis; b) subjects undergoing anti-inflammatory therapies.
  Interventions: Genetic: blood sample examination
- healthy controls: 51 age sex matched controls, patients with diagnosed with cataracts; of both sexes, aging more than 18 years. The exclusion criteria are: a) subjects with autoimmune diseases, tumors, kidney diseases, atherosclerosis; b) subjects undergoing anti-inflammatory therapies.
  Interventions: Genetic: blood sample examination

INTERVENTIONS:
Genetic: blood sample examination — droplet digital PCR in blood sample for research of mutations of GNA11 and GNAQ genes and the following microRNAs: miR - 506-514 cluster, hsamiR - 592 and hsa - miR - 199a - 5p.

SUMMARY:
The aim of the study is to identify genetic and epigenetic biomarkers in uveal melanoma, and to evaluate their diagnostic and prognostic role.

In particular, the specific objectives are:

1. to identify the circulating somatic mutations associated with uveal melanoma;
2. to identify the de-regulated miRNAs associated with uveal melanoma;
3. to evaluate the diagnostic and prognostic role of the identified genetic and epigenetic markers;
4. to identify possible therapeutic targets.

DETAILED DESCRIPTION:
This is a prospective, multicentric, case-control study, aimed at studying the gene and epigenetic mechanisms involved in uveal melanoma.

Patients with uveal melanoma, will be enrolled. For each subject included in the study, in a blood sample will be searched the mutations of the GNA11 and GNAQ genes and the expression of the following microRNAs: miR - 506-514 cluster, hsamiR - 592 and hsa - miR - 199a - 5p; the digital PCR droplet system will be used.

The study will not change the diagnostic-therapeutic process adopted in the clinical practice and will have no influence on the clinical management of enrolled patients.

A group of age sex matched controls will be recruited among patients scheduled for cataract surgery.

The sample size was calculated to detect, with a power of 80% and a confidence interval of 95%, a difference of 13.5% between the incidence of mutation of the GNA11 gene in patients with melanoma and healthy controls. (13.5% vs 0%). Overall, at least 51 patients with uveal melanoma and 51 controls will be recruited, for a total of at least 102 subjects.

ELIGIBILITY:
Inclusion Criteria:

* subjects diagnosed with uveal melanoma
* both sexes
* age ≥ 18 years

Exclusion Criteria:

* a) autoimmune diseases
* b) tumors
* c) kidney diseases
* d) atherosclerosis
* e) subjects undergoing anti-inflammatory therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uveal melanoma and controls will be recruited in three centers:
  1. the Ophthalmology Clinic of the "Policlinico-Vittorio Emanuele" University Hospital, Catania, Italy
  2. the Ophthalmology Clinic of the University of Turin, Italy
  3. the Department of General and Pediatric Ophthalmology, Medical University of Lublin, Lublin, Poland
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
circulating GNA11 mutation detection through digital droplet PCR | at the diagnosis of uveal melanoma (first visit), through study completion, in an average of 1 year
  the incidence of GNA11 mutations in uveal melanoma patients and in controls

SECONDARY OUTCOMES:
micro RNA levels in serum | at the diagnosis of uveal melanoma (first visit), through study completion, in an average of 1 year
  the expression levels of circulating miRNAs (miR - 506-514 cluster, hsamiR - 592 and hsa - miR - 199a - 5p) in uveal melanoma patients and in controls

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (2):
  - Eye Clinic, Azienda Policlinico San Marco, Catania
  - Eye Clinic University of Turin, Turin
- Department of General and Pediatric Ophthalmology, Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krantz BA, Dave N, Komatsubara KM, Marr BP, Carvajal RD. Uveal melanoma: epidemiology, etiology, and treatment of primary disease. Clin Ophthalmol. 2017 Jan 31;11:279-289. doi: 10.2147/OPTH.S89591. eCollection 2017. PMID 28203054
- [Background] Diener-West M, Reynolds SM, Agugliaro DJ, Caldwell R, Cumming K, Earle JD, Hawkins BS, Hayman JA, Jaiyesimi I, Jampol LM, Kirkwood JM, Koh WJ, Robertson DM, Shaw JM, Straatsma BR, Thoma J; Collaborative Ocular Melanoma Study Group. Development of metastatic disease after enrollment in the COMS trials for treatment of choroidal melanoma: Collaborative Ocular Melanoma Study Group Report No. 26. Arch Ophthalmol. 2005 Dec;123(12):1639-43. doi: 10.1001/archopht.123.12.1639. PMID 16344433
- [Background] Van Raamsdonk CD, Griewank KG, Crosby MB, Garrido MC, Vemula S, Wiesner T, Obenauf AC, Wackernagel W, Green G, Bouvier N, Sozen MM, Baimukanova G, Roy R, Heguy A, Dolgalev I, Khanin R, Busam K, Speicher MR, O'Brien J, Bastian BC. Mutations in GNA11 in uveal melanoma. N Engl J Med. 2010 Dec 2;363(23):2191-9. doi: 10.1056/NEJMoa1000584. Epub 2010 Nov 17. PMID 21083380
- [Background] Falzone L, Romano GL, Salemi R, Bucolo C, Tomasello B, Lupo G, Anfuso CD, Spandidos DA, Libra M, Candido S. Prognostic significance of deregulated microRNAs in uveal melanomas. Mol Med Rep. 2019 Apr;19(4):2599-2610. doi: 10.3892/mmr.2019.9949. Epub 2019 Feb 11. PMID 30816460